CLINICAL TRIAL: NCT05797740
Title: Cladribine Tablets Level of Response Predictors in Clinical Practice (CLODINA)
Status: Active, not recruiting | Type: Observational
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: MS700568_0213
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Relapsing Multiple Sclerosis; Mavenclad; Cladribine Tablets
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cladribine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single cohort: This is a single cohort study enrolling Participants with relapsing multiple sclerosis (RMS), who are prescribed treatment with cladribine tablets in routine clinical practice following the summary of product characteristics (SmPC).
  Interventions: Drug: Mavenclad

INTERVENTIONS:
Drug: Mavenclad — This is an observational study, participants who received cladribine tablets in routine clinical practice following the SmPC will be included.
  Other Names: Cladribine

SUMMARY:
This study aims to describe participants characteristics that can predict the safety and effectiveness of cladribine tablets, as assessed by time-to-discontinuation of treatment with cladribine tablets, and to assess other patient-reported, clinical, and imaging outcomes in participants with relapsing multiple sclerosis (RMS) in the long term, in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, male or female patients ≥ 18 years old at index date
* Participants must voluntarily give written informed consent form (ICF). Patients must read and fully understand the ICF
* Participants with confirmed diagnosis of RMS at index date, diagnosed by the treating physician according to applicable clinical practice guidelines (currently McDonald 2017 criteria), with high disease activity.
* Required historical data should be available: number of relapses in the 12 months prior to index date, DMTs taken prior to index date, date of MS diagnosis, and data of at least 1 MRI prior to index date as specified in the drug Summary of Product Characteristics (SmPC)
* Fulfillment of the indication for treatment with cladribine tablets at index date, per standard of care in accordance with the local SmPC
* Meeting 1 of the following criteria:

  * Prospective participants: Having been prescribed with cladribine tablets or having taken at least one dose of cladribine tablets, with enrollment date prior to the second treatment week
  * Retrospective participants: Having taken at least one dose of cladribine tablets, with enrollment date during or after the second treatment week but not more than 3 years after the first dose of cladribine tablets

Exclusion Criteria:

* Contraindications to use of cladribine tablets according to the SmPC.
* Any participant who had the first dose of cladribine tablets more than 3 years prior to enrollment
* Any participant who is pregnant or plans to breast-feed while taking cladribine tablets, or any patient who or whose partner plans to become pregnant in Year 1 or within 6 months after the last dose in Year 2, or any participants who is unwilling or unable to use contraception per the SmPC
* Have participated or participating in an interventional study since cladribine tablet initiation, in which participant assessment and/or treatment may be dictated by a protocol
* Participants who, at the discretion of the Investigator, will not be able to provide reliable information for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolls participants with a confirmed diagnosis of RMS (with high disease activity) who have been prescribed, have initiated, or have completed/discontinued treatment with cladribine tablets per the decision of the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Time to Discontinuation of Treatment with Cladribine tablets | Up to 48 months

SECONDARY OUTCOMES:
Percentage of participants Receiving Each of The Possible Number of Annual Treatment Courses with Cladribine Tablets | Baseline, 12 months, 24 months, 36 months and 48 months
Cumulative Cladribine Dose | Up to 48 months
Number of Relapses | Baseline, 12 months, 24 months, 36 months and 48 months
Proportion of Severe Relapses | Baseline, 12 months, 24 months, 36 months and 48 months
Percentage of Participants Free From Relapse | Year 2 and Year 4
Time From Onset of Relapse to Recovery | Up to Month 48
Annualized Relapse Rate (ARR) | At Year 2 and Year 4
Percentage of Participants Free From Magnetic Resonance Imaging (MRI) Activity | At Year 1, Year 2, Year 3 and Year 4
Percentage of Participants with Minimal MRI Activity (=< 2 New T2 Lesions) | At Year 1, Year 2, Year 3 and Year 4
Timed 25-Foot Walk (T25FW) Score | Baseline, Year 1, Year 2, Year 3 and Year 4
Percentage of Participants with an Increase and Decrease in Timed 25-Foot Walk (T25FW) Score of At Least 20% From Baseline at Year 1, 2, 3 and 4 | Baseline, Year 1, Year 2, Year 3 and Year 4
9-Hole Peg Test (9HPT) Score | Baseline, Year 1, Year 2, Year 3 and Year 4
Percentage of Participants with an Increase and Decrease in 9-Hole Peg Test (9HPT) Score of At Least 20% From Baseline at Year 1, 2, 3 and 4 | Baseline, Year 1, Year 2, Year 3 and Year 4
Percentage of Participants With Progressed, Improved, or Stable Disability as Assessed by Expanded Disability Status Scale (EDSS) Confirmed Over 6 Months | Year 1, Year 2, Year 3 and Year 4
Percentage of Participants With Sustained Disability Progression, Improvement, or Stability Confirmed Over 6 Months as Assessed by T25FW Score | Year 1, Year 2, Year 3 and Year 4
Percentage of Participants With Sustained Disability Progression, Improvement, or Stability Confirmed Over 6 Months as Assessed by 9HPT Score | Year 1, Year 2, Year 3 and Year 4
Percentage of Participants With Minimal Evidence of Disease Activity (MEDA) | Year 2 and Year 4
Percentage of Participants With No Evidence of Disease Activity (NEDA-3) | Year 2 and Year 4
Multiple Sclerosis Impact Scale (MSIS-29) Physical Domain Score, Psychological Domain Score and Total Score | Baseline, Year 1, Year 2, Year 3 and Year 4
EuroQol 5-Dimensions (EQ-5D-5L) Score | Baseline, Year 1, Year 2, Year 3 and Year 4
Global Satisfaction, Effectiveness, Side Effects, and Convenience Domain Scores of Treatment Satisfaction Questionnaire for Medication (TSQM) | Baseline, Year 1, Year 2, Year 3 and Year 4
Treatment Cost of Disease-Modifying Treatment (DMTs) | Up to 48 months
EuroQol Visual Analog Scale (EQ-VAS) Score | Baseline, Year 1, Year 2, Year 3 and Year 4

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (30):
- Belgium (4):
  - UCL Saint Luc, Brussels
  - UZ Antwerpen, Edegem
  - AZ Groeninge vzw, Kortrijk
  - CHU Sart Tilman, Liège
- Czechia (5):
  - FN u sv. Anny Brno, Brno
  - FN Hradec Králové, Hradec Králové
  - NeuropsychiatrieHK, Hradec Králové
  - Fakultni nemocnice Ostrava, Ostrava
  - Nemocnice Teplice, Teplice
- Greece (13):
  - University of Thrace, Medical School - Neurology Department, Alexandroupoli, Alexandroupoli
  - Aiginiteio' Hospital, Athens
  - Attikon, Athens
  - Evagelismos, Athens
  - General Miliary Hospital of Athens "401", Athens
  - University of Ioannina - Neurology department, Ioannina
  - University Hospital of Larissa, Larissa
  - General Hospital "Agios Andreas", Pátrai
  - University of Patras, Pátrai
  - AHEPA University Hospital of Thessaloniki, Thessaloniki
  - General Hospital of Athens G.Gennimatas, Thessaloniki
  - Interbalkan Hospital of Thessaloniki, Thessaloniki
  - St Luke's Clinic, Thessaloniki
- Zuyderland, Sittard-Geleen, Netherlands
- Poland (3):
  - Oddział Kliniczny Neurologii, Szpital Uniwersytecki w Krakowie, Krakow
  - Medical Academy Neurology Clinic, Poznan
  - Szpital Kliniczny Nr 1 Pomorskiego Uniwersytetu Medycznego w Szczecinie, Szczecin
- Portugal (4):
  - Centro Hospitalar e Universitario de Coimbra, Coimbra
  - Centro Hospitalar Lisboa Norte Hospital de Santa Maria, Lisbon
  - Centro Hospitalar Universitário Lisboa Central - Hospital dos Capuchos, Lisbon
  - Centro Hospitalar de São João E. P. E., Porto

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS700568_0213
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html